CLINICAL TRIAL: NCT03219658
Title: STOMP Early Years: A Pilot Randomized Controlled Trial of an Intensive, Family-Centred, Home Visiting Intervention for Young Children With Severe Obesity
Brief Title: STOMP Early Years: A Pilot RCT of an Intensive, Family-Centred, Home Visiting Intervention for Young Children With Severe Obesity
Acronym: STOMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Catherine Birken, Staff Paediatrician, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1000054922
Record Dates: First submitted 2017-06-27; First posted 2017-07-17 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Child Obesity
Keywords: Parenting; Home visiting; Childhood obesity treatment
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parenting education sessions (Experimental): Receive 10 weeks of group parenting education sessions with 2-4 public health nurse home visits.
  Interventions: Behavioral: Parenting education sessions
- Control (No Intervention): Attend one-on-one check-ins with the interdisciplinary team at STOMP; wait-listed control group.

INTERVENTIONS:
Behavioral: Parenting education sessions — If assigned to the parenting education session group, families will start with the 10-week group parenting education sessions and 2-4 home visits immediately after being enrolled. During this time, they will also come in for four one-on-one check-ins with the STOMP team. Each check-in will be approximately 1 hour. At least one parent/caregiver will attend weekly parenting sessions which will take place at SickKids. The Toronto Public Health Nurse will arrange 2-4 home visits with the family during the 6 month period of the study. The home visits will focus on helping to apply the messages and skills from the group sessions in their homes, and making connections in the neighbourhood to recreational or nutrition programs or other supports for the family.
  Arms: Parenting education sessions

SUMMARY:
This internal pilot study will determine whether a highly promising primary care based intervention that combines group based parenting skills training and public health nurse home visits with a focus on healthy nutrition, activity and sleep, will lead to improved weight status in 1 to 5 year old children with severe obesity.

Children with severe obesity will be identified through the obesity management clinical program at The Hospital for Sick Children called STOMP (SickKids Team Obesity Management Program). The STOMP Early Years Program is a unique and intensive, paediatric obesity management program designed for 1 to 5 year-olds with severe obesity and their families. Families who participate in this study will be randomly assigned (having an equal chance of being in either group) to one of the two study groups that will run for 6 months:

Group A: Ten weeks of group parenting education sessions with 2-4 public health nurse home visits and four one-on-one check-ins with an interdisciplinary team at STOMP.

Group B: Wait listed to receive parenting education sessions; receive one-on-one checks with an interdisciplinary team at STOMP.

In addition to the measures collected as part of STOMP, families will complete the following questionnaires before the start of the trial, and after 6 months:

Parenting Scale, Parenting Stress Index, Depression, Anxiety, and Stress Scale (DASS-21), Cost Questionnaire, and Children's Behaviour Questionnaire (CBQ).

ELIGIBILITY:
Inclusion Criteria:

* Children with obesity and severe obesity (BMI ≥97th percentile) and at least one parent (primary caregiver), and families who are fluent in English (written and oral) will be eligible to participate.

Exclusion Criteria:

* Children with diagnosed Prader-Willi syndrome; severe developmental delay; and families who reside beyond the Toronto Public Health catchment area for home visiting.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
zBMI | 6 months post-intervention
  Measure the difference in age and sex-standardized BMI z-score (zBMI)

SECONDARY OUTCOMES:
Mental health | 6 months post-intervention
  Assess mental health by Strengths and Difficulties Questionnaire
Eating behaviour and dietary intake | 6 months post-intervention
  Assess eating behaviour and dietary intake using the Nutrition Screening Tool for Every Preschooler (NutriSTEP)

OTHER OUTCOMES:
Parent report focus group | 6 months post-intervention
  focus group of eligible parents around feasibility and acceptability of the planned intervention

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kinlin LM, Oreskovich SM, Dubrowski R, Ball GDC, Barwick M, Dettmer E, Haines J, Hamilton J, Kim THM, Klaassen M, Luca P, Maguire JL, Moretti ME, Stasiulis E, Toulany A, Birken CS. Managing Obesity in Young Children: A Multiple Methods Study Assessing Feasibility, Acceptability, and Implementation of a Multicomponent, Family-Based Intervention. Child Obes. 2022 Sep;18(6):409-421. doi: 10.1089/chi.2021.0221. Epub 2022 Jan 26. PMID 35085455